CLINICAL TRIAL: NCT02680275
Title: Efficacy of Intravaginal Dead Sea Peloid Gel Administration in Complex Treatment of Chronic Endometritis and Reproductive Disorders: Randomized Placebo-controlled Prospective Study
Brief Title: Efficacy of Dead Sea Peloid Gel in Chronic Endometritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scientific Center for Family Health and Human Reproduction Problems, Russia (Other Government)
Responsible Party: Principal Investigator, Irina N. Danusevich, Principal Investigator, Scientific Center for Family Health and Human Reproduction Problems, Russia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16
Record Dates: First submitted 2015-12-22; First posted 2016-02-11 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2015-09

CONDITIONS: Chronic Endometritis
Keywords: Chronic endometritis; Miscarriage; Infertility
MeSH Terms: conditions — Abortion, Spontaneous; Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Doxycycline,Dead Sea Peloid Gel,placebo (Experimental): 1. Group -1 stage: Doxycycline 100mg 2 times per day 10 days; followed by Dead Sea Peloid Gel , 60 ml per day fo 12 days, intravaginally
  2. Group -1 stage: Doxycycline 100mg 2 times per day 10 days; followed by placebo gel, 60 ml per day fo 12 days, intravaginally
  Interventions: Drug: Dead Sea Peloid Gel

INTERVENTIONS:
Drug: Dead Sea Peloid Gel — intravaginally
  Other Names: Placebo Gel

SUMMARY:
This study evaluates the effect of Dead Sea Peloid Gel in the treatment of Chronic Endometritis in women with reproductive disorders. Half of participants will receive Dead Sea Peloid Gel and antibiotics, while the other half will receive Placebo Gel and antibiotics.

Patients with reproductive disorders who visited Research Medical Center of Family Health Problems and Human Reproduction were recruited.

DETAILED DESCRIPTION:
Dead Sea Peloid Gel achieves improvement of blood circulation and receptor sensitivity of endometrium.

ELIGIBILITY:
Inclusion Criteria:

* Women with miscarriage associated with chronic endometritis
* Women without mental disorders able to swallow tablets

Exclusion Criteria: Clinical diagnosis of:

* sexually transmitted diseases
* endometrium hyperplasia and/or polyps
* uterina fibroids
* endocrine disorders
* trombophilia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The prevalence of spontaneous pregnancy the first year after treatment | during first year

SECONDARY OUTCOMES:
The prevalence of women with morphological status of chronic endometritis by the 3 months after treatment. | during 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Marina A Darenskaya, MD, Study Chair — Scientific Center for Family Health and Human Reproduction Problems
Locations (1):
- Scientific Center for Family Health and Human Reproduction Problems, Irkutsk, Russia

IPD SHARING:
Plan to Share IPD: No
The study can generate the publications related to the outcomes. The investigator initiating the protocol (Protocol leader/coPI) will be the first (primary) author of the publication. The publication wil also could involve the names of the site investigators who have contributed to the study. The authorship order of the site investigators will be based upon personal contribution to the study, approved by the SCFHHRP (sponsor). The primary affiliation of the study is SCFHHRP.